CLINICAL TRIAL: NCT04340947
Title: Impact of a Reduced Nicotine Standard on Young Adult Appeal for Menthol and Non-menthol Cigarettes
Brief Title: Cigarette Smoking Among Young Adults
Acronym: ENHANCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: ENHANCE; R01DA050990 (NIH)
Record Dates: First submitted 2020-03-25; First posted 2020-04-10 (Actual); Results first posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Cigarette Smoking; Smoking Behaviors
MeSH Terms: conditions — Cigarette Smoking; Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Menthol very low nicotine cigarette (VLNC), then non-menthol VLNC (Experimental): Participants will smoke menthol flavored very low nicotine cigarettes in their home environment for 7 days. At the end of 7-days, they will also smoke one menthol flavored very low nicotine cigarette in the laboratory.
  Interventions: Other: Very low nicotine cigarette: menthol; Other: Very low nicotine cigarette: non-mentol
- Non-menthol very low nicotine cigarette (VLNC), then menthol VLNC (Experimental): Participants will smoke non-menthol flavored very low nicotine cigarettes in their home environment for 7 days. At the end of 7-days, they will also smoke one non-menthol flavored very low nicotine cigarette in the laboratory.
  Interventions: Other: Very low nicotine cigarette: menthol; Other: Very low nicotine cigarette: non-mentol

INTERVENTIONS:
Other: Very low nicotine cigarette: menthol — Participants will be randomized to smoke either menthol non-menthol flavored very low nicotine cigarettes in their home environment for 7 days and in the laboratory first and then crossed over to receive the opposite intervention. The study consists of two treatment periods of 7 days separated by a 1 week wash-out period
Other: Very low nicotine cigarette: non-mentol — Participants will be randomized to smoke either menthol non-menthol flavored very low nicotine cigarettes in their home environment for 7 days and in the laboratory first and then crossed over to receive the opposite intervention. The study consists of two treatment periods of 7 days separated by a 1 week wash-out period

SUMMARY:
This study will examine perceptions and smoking behavior of menthol and non-menthol very low nicotine cigarettes in young adult smokers. The aims are to examine perceptions and smoking behavior in the laboratory and in the natural environment. A separate sub-sample of men and women who identify as LGBTQ2S+ will also be recruited.

DETAILED DESCRIPTION:
This proposal includes three different aspects of assessment for menthol smoking young adults. The laboratory phase includes three separate sessions of laboratory smoking through a machine designed to measure puff behavior; the EMA phase includes 21 days of monitoring smoking behavior and attitudes related to smoking when smoking one's usual brand cigarette, the assigned menthol low nicotine cigarette, and the assigned non-menthol low nicotine cigarette in the participant's natural environment. The order of administration of smoking menthol and non-menthol VLNC will be counterbalanced. There will be a 7-day wash-out period between each 7-day period of using low nicotine cigarettes. The final phase includes a virtual marketplace where participants can purchase and use the research cigarettes in the context of other available tobacco products on the market, or purchase no tobacco products at all. There will be a final assessment, over the phone or in-person, 30-days after the final study visit (at week 8), to assess tobacco use behavior and attitudes about tobacco use. Participants will be enrolled for approximately 9 weeks. Week 1 will consist of smoking one's usual brand of cigarette in the laboratory and then in their home environment for 7-days. Week 2 will consist of smoking the first very low nicotine cigarette in the home environment for 7 days and then in the laboratory. Week three will consist of a 7-day wash-out period where participants can smoke their usual brand again, as they normally would. Week 4 will consist of smoking the second very low nicotine cigarette at home for 7 days and then in the laboratory. Week 5 will consist of returning to the laboratory for a final study visit and complete a hypothetical experimental tobacco marketplace. One month (4 weeks) after the final study visit (week 9), participants will complete a 30-day follow-up of cigarette smoking and other tobacco use behavior.

ELIGIBILITY:
Inclusion Criteria:

1. Ages18 to 34;
2. Smoke cigarettes "somedays" or "everyday" for at least the past 3-months;
3. A strong preference for menthol cigarettes (i.e., smoke menthol >80% of the time); and
4. Ability to read English at an 8th grade level or higher;
5. No immediate plans to quit smoking.

Exclusion Criteria:

1. Current use of nicotine replacement therapy (NRT);
2. Pregnant or planning to become pregnant, or currently breastfeeding;
3. Past or current self-reported clinically significant heart disease or hypertension, or other smoking-related disease (by history) that preclude successful study completion;
4. Serious psychiatric disorder;
5. Inability to abstain from nicotine/tobacco products;
6. Strong preference for non-menthol cigarettes (smoke non-menthol > 80% of the time)

Ages: 18 Years to 34 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 171 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy Cohn, PhD, Principal Investigator — University of Oklahoma
Locations (1):
- Health Promotion Research Center, Oklahoma City, Oklahoma, United States

REFERENCES:
- [Derived] Cohn AM, Cassidy R, Denlinger-Apte R, Donny E, Villanti AC, Hatsukami D, Dunn D, Wyatt R, Niznik T, Cohen-Davidyan T, Smith M, Ehlke SJ. Impact of a reduced nicotine standard on young adult appeal for menthol and non-menthol cigarettes. BMJ Open. 2022 Nov 21;12(11):e067694. doi: 10.1136/bmjopen-2022-067694. PMID 36410805

RESULTS

PARTICIPANT FLOW:
Recruitment Details: N= 171 were eligible and enrolled at the first visit. N=143 people attended Visit 2 to smoke their usual brand (UB) cigarette, and n=139 were randomized to the intervention. After visit 2, the intervention began where people smoked a menthol and non-menthol VLNC (order counterbalanced) in two subsequent visits (VLNC 1 visit, VLNC 2 visit). There was a 7-day washout period between VLNC 1 and VLNC 2 smoking. The experimental tobacco marketplace was the final visit.
Pre-assignment Details: This is a within-subjects design. Participants were assigned to both smoke menthol and non-menthol very low nicotine cigarettes in visits 3 and 4 and at home for a week prior to each visit. The order of administration of menthol vs non-menthol flavor was counterbalanced to reduce the impact of order effects. The number of people to start a period may not equal the number who completed the previous period due to loss to follow-up.
Groups:
- Menthol Very Low Nicotine Cigarette First; Non-menthol Very Low Nicotine Cigarette First: Participants complete a within-subject design where they smoke both a menthol and a non-menthol very low nicotine cigarette; the order of administration of menthol vs non-menthol very low nicotine cigarette smoking is counterbalanced.
Period: Usual Brand Smoking (Visit 2)
Arm/Group | Menthol Very Low Nicotine Cigarette First | Non-menthol Very Low Nicotine Cigarette First
Started | 69 | 70
Completed | 69 | 70
Not Completed | 0 | 0
Period: VLNC 1 Smoking (Visit 3)
Arm/Group | Menthol Very Low Nicotine Cigarette First | Non-menthol Very Low Nicotine Cigarette First
Started | 56 (People who attended the first VLNC smoking visit) | 60 (People who attended the first VLNC smoking visit)
Completed | 56 | 60
Not Completed | 0 | 0
Period: 7-day Washout Period
Arm/Group | Menthol Very Low Nicotine Cigarette First | Non-menthol Very Low Nicotine Cigarette First
Started (People who started the 7-day washout period) | 56 | 60
Completed | 51 | 56
Not Completed | 5 | 4
Not completed — Lost to Follow-up | 5 | 4
Period: VLNC 2 Smoking (Visit 4)
Arm/Group | Menthol Very Low Nicotine Cigarette First | Non-menthol Very Low Nicotine Cigarette First
Started | 51 (People who attended the second VLNC smoking visit) | 56 (People who attended the second VLNC smoking visit)
Completed | 51 | 56
Not Completed | 0 | 0
Period: Experimental Tobacco Marketplace (Visit)
Arm/Group | Menthol Very Low Nicotine Cigarette First | Non-menthol Very Low Nicotine Cigarette First
Started | 49 (People who attended the final study visit) | 54 (People who attended the final study visit)
Completed | 49 | 54
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: N=171 participants completed the baseline visit and were eligible at the end of that visit
Groups:
- All Study Participants: Participants will smoke menthol flavored very low nicotine cigarettes in their home environment for 7 days. At the end of 7-days, they will also smoke one menthol flavored very low nicotine cigarette in the laboratory.
  Very low nicotine cigarettes: Participants were randomized to smoke menthol and non-menthol flavored very low nicotine cigarettes in their home environment for 7 days and in the laboratory.
Arm/Group | All Study Participants
Number analyzed (Participants) | 171
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.16 (4.41)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Data on sex missing for 1 person.
  Participants
    Female | 84
    Male | 87
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Data missing on 1 participant
  Participants
    Non-hispanic Black | 22
    Non-hispanic white | 102
    Non-hispanic other race | 25
    Hispanic | 22
Region of Enrollment [Number; unit: participants]
  United States | 171
Cigarettes/day [Mean (Standard Deviation); unit: unit of measure "cigarettes per day"] — Number of cigarettes smoked per day
  unit of measure "cigarettes per day" | 8.86 (6.58)
Time-to-first cigarette [Count of Participants; unit: Participants] — Population: Data missing for n=1
  Participants
    Smoke within 5 minutes of waking: number analyzed (Participants) | 170
    Smoke within 5 minutes of waking | 36
    Smoke within 6 or more minutes after waking: number analyzed (Participants) | 170
    Smoke within 6 or more minutes after waking | 134

OUTCOME MEASURES:

1. Primary Outcome: Puff Topography
Description: total inhalation volume from smoking behavior in the laboratory
Time Frame: Baseline to week 4
Population: Analysis was restricted to individuals who completed at 2 study visits (of 3 visits). Some individuals were excluded from analysis because of missing smoking data that was not captured by the smoking topography device or several participants who erroneously smoked more than 1 cigarette.
Measure: Mean (Standard Deviation); unit: mL
Groups:
- Usual Brand Cigarette: After baseline, participants are instructed to smoke their usual brand as they would for 7 days and then return to the laboratory and smoke 1 of their usual brand cigarettes in the lab. Participants are then randomly assigned, through counterbalancing, to smoke a menthol very low nicotine and a non-menthol very low nicotine cigarette (order counterbalanced) in the following visits 3 and 4.
- Menthol Very Low Nicotine Cigarette; Non-menthol Very Low Nicotine Cigarette: Participants complete a within-subject design where they smoke both a menthol and a non-menthol very low nicotine cigarette; the order of administration of menthol vs non-menthol very low nicotine cigarette smoking is counterbalanced.
Arm/Group | Usual Brand Cigarette | Menthol Very Low Nicotine Cigarette | Non-menthol Very Low Nicotine Cigarette
Number analyzed (Participants) | 111 | 99 | 103
mL | 1108 (1013.7) | 1045.2 (1119.4) | 1084.6 (1141)

2. Primary Outcome: Ratings of Psychological Reward
Description: Subjective response to smoking, as measured by self-reported psychological reward (scale) of the modified Cigarette Evaluation Scale, administered after smoking. The minimum value is 1 and the maximum value is 7; with 7 indicating greater psychological reward.
Time Frame: Baseline to week 9
Population: Population included participants who completed at two study visits and who did not have any missing data on the outcomes
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Brand Cigarette | Menthol Very Low Nicotine Cigarette | Non-menthol Very Low Nicotine Cigarette
Number analyzed (Participants) | 111 | 111 | 111
score on a scale | 3.1 (1.30) | 2.9 (1.40) | 2.3 (1.30)

3. Primary Outcome: Hypothetical Purchasing of Non-Menthol Very Low Nicotine Cigarettes (VLNCs)
Description: Purchasing of non-menthol very low nicotine cigarettes in the Experimental Tobacco Marketplace (ETM) task 1 and 2. Product units purchased per cigarette price displayed in the ETM, displayed as milligrams of nicotine. Prices are $0.12, $0.25, $0.5, $1, $2, $4, $8, and $16 per cigarette. Data are presented as units purchased on a log scale, per recommended best practices.
Time Frame: Assessed during tobacco purchase tasks completed at week 5
Population: We report raw data on number of non-menthol VLNCs purchased at each price.
Measure: Mean (Standard Deviation); unit: log (mg of nicotine)
Groups:
- Experimental Tobacco Marketplace 1: Participants completed 2 experimental tobacco marketplace (ETM) tasks at visit 5, the final study visit. ETM 1 assessed desire to purchase non-menthol very low nicotine cigarettes (displayed as milligrams of nicotine) at 8 escalating prices.
- Experimental Tobacco Marketplace 2: Participants completed 2 experimental tobacco marketplace (ETM) tasks at visit 5, the final study visit. ETM 2 assessed desire to purchase non-menthol and non-menthol very low nicotine cigarettes (displayed as milligrams of nicotine) at 8 escalating prices.
Arm/Group | Experimental Tobacco Marketplace 1 | Experimental Tobacco Marketplace 2
Number analyzed (Participants) | 103 | 103
log (mg of nicotine)
  $0.12 | 20.40 (36.22) | 6.11 (18.38)
  $0.25 | 14.44 (26.64) | 3.66 (13.11)
  $0.50 | 10.17 (19.25) | 3.37 (12.21)
  $1.00 | 5.68 (14.64) | 1.68 (7.21)
  $2.00 | 2.56 (7.56) | 1.18 (6.33)
  $4.00 | 1.16 (6.04) | 0.34 (1.69)
  $8.00 | 0.44 (2.13) | 0.06 (0.43)
  $16.00 | 0.25 (1.51) | 0.02 (0.13)

4. Secondary Outcome: Exhaled CO Boost
Description: measures expired alveolar carbon monoxide (CO) level before smoking and after smoking; measured in parts per million (ppm)
Time Frame: Baseline to week 4
Population: Population included individuals who completed at least 2 study visits and who did not have any missing data.
Measure: Mean (Standard Deviation); unit: parts per million (ppm)
Arm/Group | Usual Brand Cigarette | Menthol Very Low Nicotine Cigarette | Non-menthol Very Low Nicotine Cigarette
Number analyzed (Participants) | 92 | 92 | 92
parts per million (ppm)
  Before smoking | 4.08 (5.03) | 3.72 (4.16) | 3.9 (5.12)
  After smoking | 9.17 (9.42) | 7.65 (6.84) | 6.79 (6.80)

5. Other Pre Specified Outcome: Nicotine Withdrawal
Description: Symptoms of nicotine withdrawal were measured using the Minnesota Nicotine Withdrawal Scale. Response options range from 0=none to 4=severe; where higher scores indicate more severe nicotine withdrawal.
Time Frame: Baseline to week 9
Population: Population included individuals who completed at least 2 study visits and who did not have any missing data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Brand Cigarette | Menthol Very Low Nicotine Cigarette | Non-menthol Very Low Nicotine Cigarette
Number analyzed (Participants) | 92 | 92 | 92
score on a scale
  Before smoking | 0.54 (0.47) | 0.48 (.41) | 0.47 (0.45)
  After smoking | .26 (.29) | .27 (.30) | .30 (.29)

6. Other Pre Specified Outcome: Change in Cigarette Craving Before and After Smoking
Description: 1-item craving measure from the Minnesota Nicotine Withdrawal Scale. Response options range from 0 (none/not at all) to 4 (severe), where 4 indicates higher craving for a cigarette.
Time Frame: Baseline to week 9
Population: Population included individuals who completed at least 2 study visits and who did not have any missing data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Brand Cigarette | Menthol Very Low Nicotine Cigarette | Non-menthol Very Low Nicotine Cigarette
Number analyzed (Participants) | 92 | 92 | 92
score on a scale | 2.18 (1.38) | 1.92 (1.43) | 1.85 (1.33)

7. Other Pre Specified Outcome: Perceived Health Risk Scale
Description: This scale measures perceptions of risk from smoking one's usual brand or the very low nicotine cigarettes. Participants completed this questionnaire at the beginning of each in-person smoking visit (after a week of smoking the assigned cigarette at home). The measure has 7 questions. Each question has response options ranging from 1 (very low risk of disease) to 10 (very high risk of disease). Higher scores indicate greater perceived risk. The outcome reflects the total score, divided by 7 (the number of questions)
Time Frame: Baseline to week 8
Population: Population includes individuals who attended the visit and who completed the questionnaire on perceived health risks of the cigarette flavor they smoked in the previous week.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Brand Cigarette | Menthol Very Low Nicotine Cigarette | Non-menthol Very Low Nicotine Cigarette
Number analyzed (Participants) | 135 | 111 | 107
units on a scale | 5.30 (2.2) | 4.45 (2.28) | 4.45 (2.18)

8. Other Pre Specified Outcome: Heart Rate
Description: Heart rate is measured as beats per minute (BPM); where higher scores indicate higher heart rate.
Time Frame: Baseline to week 4
Population: Population included individuals who completed at least 2 study visits and who did not have any missing data.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Usual Brand Cigarette | Menthol Very Low Nicotine Cigarette | Non-menthol Very Low Nicotine Cigarette
Number analyzed (Participants) | 92 | 92 | 92
beats per minute
  Before smoking | 76.85 (12.38) | 75.03 (13.62) | 77.25 (12.77)
  After smoking | 85.73 (14.06) | 75.72 (14.38) | 76.42 (13.00)

ADVERSE EVENTS:
Time Frame: 4 months
Description: The definition does not differ. Adverse events were collected via a self-report form at the beginning of each in person visit.
Groups:
- All Participants: All participants enrolled in the study, n=171
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/171
Serious Adverse Events (participants affected / at risk) | 0/171
Other Adverse Events (participants affected / at risk) | 1/171
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=171)
Respiratory symptoms (Respiratory, thoracic and mediastinal disorders) | 1 (1) — At second study session, participant reported heart palpitations on the Adverse Events forms, prior to smoking their usual cigarette. All vitals were within range. The participant was withdrawn from the study for safety concerns.

LIMITATIONS AND CAVEATS:
We focused on young adults who smoke menthol cigarettes. Findings may not generalize to non-menthol smokers or to different age groups. We did not include menthol and non-menthol normal nicotine cigarette conditions. Participants were not blinded to the cigarette nicotine content to model real-world conditions where consumers are aware of the cigarettes they smoke.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-11-16): https://cdn.clinicaltrials.gov/large-docs/47/NCT04340947/Prot_SAP_000.pdf